CLINICAL TRIAL: NCT04245319
Title: Assessment of the Combined Effect of Acitretin and Narrow Band Ultraviolet B (Nb-UVB) on the Clinical Repigmentation and on the Expression of E-cadherins in Vitiligo Lesions in Comparison to Narrow Band UVB Alone. A Pilot Study
Brief Title: Combined Effect of Acitretin and Narrow Band Ultraviolet B on Vitiligo Repigmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shahira Ramadan, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Acitretin in vitiligo
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Hyperlipidemias; Xerosis; Depression; Liver Diseases
MeSH Terms: conditions — Hyperlipidemias; Depression; Liver Diseases | interventions — Acitretin; Capsules

STUDY DESIGN:
Intervention Model Description: Two groups Group A: patients will receive three NB-UVB sessions per week for 48 sessions. Group B: patients will receive three NB-UVB sessions per week for 48 sessions combined with acitretin in a dose of 0.3 mg/kg/day daily.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NbUVB (Other): Group A: patients will receive three NB-UVB sessions per week for 48 sessions.
  Interventions: Other: Narrow band ultraviolet B
- Combined nbUVB and Acitretin (Experimental): Group B: patients will receive three NB-UVB sessions per week for 48 sessions combined with acitretin in a dose of 0.3mg/kg/day daily.
  Interventions: Drug: Acitretin; Other: Narrow band ultraviolet B

INTERVENTIONS:
Drug: Acitretin — The patients will receive the drug and the effect on repigmentation on vitiligo lesions will be observed
  Other Names: Acitretin 25Mg Cap; Acitretin 10Mg Cap
  Arms: Combined nbUVB and Acitretin
Other: Narrow band ultraviolet B — Patients receive nbUVB session 3 times per week

SUMMARY:
Since abnormal keratinocyte (KC) proliferation and differentiation as well as defective E cadherin expression were reported in vitiligo lesions, the investigators set to study the potential efficacy of combining Retinoids, which are known to improve KC proliferation and differentiation and increase the expression of adhesion molecules, with narrowband UVB in the treatment of vitiligo.

DETAILED DESCRIPTION:
• Twenty patients with generalized vitiligo will be included in this study.

All patients will be subjected to:

* Clinical evaluation:
* An informed written consent.
* History taking include age, previous treatment, disease activity
* Clinical examination including Vitiligo Area Scoring Index (VASI) and Vitiligo Disease Activity Score (VIDA)
* Photography (before starting the treatment and every 2 weeks till the end of the study)

Laboratory evaluation:

* 2 mm punch skin biopsies will be taken from vitiligo patients, 1 from lesional and the other from perilesional skin before treatment.
* The patients will be randomly assigned to two groups:

Group A: patients will receive three NB-UVB sessions per week for 48 sessions. Group B: patients will receive three NB-UVB sessions per week for 48 sessions combined with acitretin in a dose of 0.3mg/kg/day daily.

* Controls: 20 individuals age and sex matched will be biopsied from the skin of their abdominoplasty surgery.
* Another two 2 mm punch skin biopsies will be taken from lesional and perilesional skin at the onset of repigmentation if repigmentation starts before completion of the 48 treatment session or after completion of the treatment period if repigmentation does not occur.
* .All biopsies from patients and controls will be stained Immunohistochemically by anti-E cadherin antibody.

ELIGIBILITY:
Inclusion Criteria:

* Patients with generalized non-segmental vitiligo (25%-75%)
* Males, postmenopausal females and premenopausal females not planning to get pregnant during the period of treatment and after 2 years from the end of treatment.
* Age more than 18 years.

Exclusion Criteria:

* Children ˂ 18 years old
* Pregnant females
* Premenopausal females planning to get pregnant within the period of treatment or within 2 years after.
* Patients receiving treatment for vitiligo within the past 2 months.
* Patients with abnormal liver profile
* Patients with abnormal lipid profile
* Patients with associated photosensitive disorders
* Patients having associated skin diseases other than vitiligo
* Cataract and aphakia
* High cumulative dose from previous sessions of narrowband ˃ 200-300 session

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Determining whether addition of acitretin is beneficial for vitiligo patients or not using Vitiligo Area Scoring Index | 4-5 months
  The number of patients who will achieve 100%, 75% and 50% repigmentation of vitiligo lesions will be compared between group A (nbUVB) and group B (nbUVB+ acitretin) after 48 nbUVB sessions. The comparison of the 2 groups will be assessed using Vitiligo Area Scoring Index (VASI)
Determining whether addition of acitretin is beneficial for vitiligo patients or not using Vitiligo Disease Activity Score. | 4-5 months
  The number of patients who will achieve 100%, 75% and 50% repigmentation of vitiligo lesions will be compared between group A (nbUVB) and group B (nbUVB+ acitretin) after 48 nbUVB sessions. The comparison of the 2 groups will be assessed using Vitiligo Disease Activity Score (VIDA).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No